CLINICAL TRIAL: NCT04489394
Title: Prospective Follow-up Study of the Aesculap Quintex® Anterior Cervical Plating System After a Minimum of One Year
Brief Title: Quintex® Follow-up After One Year Minimum
Acronym: Quintex
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1901
Record Dates: First submitted 2020-07-24; First posted 2020-07-28 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis; Trauma; Spinal Stenosis; Deformity of Spine; Pseudoarthrosis of Spine; Cervical Spondylosis; Instability; Back
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis; Wounds and Injuries; Spinal Stenosis; Spondylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective study, not randomised, non-interventional, monocentric, investigating an intended patient cohort of 60 patients already operated on the cervical spine due to degenerative disc disease of the cervical spine down to the first thoracolumbar VBR (C2-T1), who received a Quintex plate for stabilisation

ELIGIBILITY:
Inclusion Criteria:

- all patients who received a Quintex® Anterior Cervical Plate since 2014 until approx. end 2018 (minimum Follow-up is one year) in the study center

Exclusion Criteria:

* Patient informed consent not signed
* Patients living outside a radius of 80 km around the study center

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Clinical Results measured by Neck Disability Index (NDI) | One retrospective visit, between one and approx. five years post-op.
  The NDI is designed to measure neck-specific disability. The questionnaire has 10 items to measure patient-reported disability secondary to neck pain and activities of daily living including personal care, lifting, reading, headaches, concentration, work status, driving, sleeping and recreation and patients rate their status from 0 (best) to 5 (worst imaginable). Individual item responses are summed to a total score, where 0 points indicate no activity limitations and 50 points indicate complete activity limitation.

SECONDARY OUTCOMES:
Neck and arm pain | One retrospective visit, between one and approx. five years post-op.
  Visual analogue scale for pain: The visual analogue scale (VAS) is a scale used to determine the pain intensity experienced by individuals. It consists of a line, approximately 10-15 cm in length, with the left side signifying no pain with a smiling face image and the right side signifying the worst pain ever with a frowning face image.
Patient satisfaction | One retrospective visit, between one and approx. five years post-op.
  Patient satisfaction with Outcome of surgery documented in two aspects: is the Patient satisfied (four Point scale:
  very satisfied, satisfied, unsatisfied, very unsatisfied) and would the Patient like to undergo surgery again (yes, no, not willing to say)
Quality of life measured by EQ-5D-5L | One retrospective visit, between one and approx. five years post-op.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/ depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Dysphagia assessment | One retrospective visit, between one and approx. five years post-op.
  Bazaz score: The Bazaz Dysphagia Score is one criterion used to define dysphagia; it classifies dysphagia as severe, moderate, mild, or none
Complications | One retrospective visit, between one and approx. five years post-op.
  Adverse Events and Serious Adverse Events, reoperations and revisions rates
Postoperative Need for Pain medication | One retrospective visit, between one and approx. five years post-op.
  The patient's Need for Pain Medication is measured by the WHO (World Health Organization) analgesic ladder
Radiological outcome from standard x-rays | One retrospective visit, between one and approx. five years post-op.
  Radiologically: Fusion status, plate position, pot. migration of screws and plate, radiolucent lines

CONTACTS AND LOCATIONS:
Locations (1):
- Katholisches Klinikum Koblenz, Koblenz, Germany

REFERENCES:
- [Result] Bruchmann B, Kilian F. Follow-up of a new titanium cervical plate for fusion of the cervical spine. Orthop Rev (Pavia). 2023 Oct 12;15:84651. doi: 10.52965/001c.84651. eCollection 2023. PMID 37842541